CLINICAL TRIAL: NCT01969786
Title: Village Integrated Eye Workers Trial
Acronym: VIEW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Eye Institute (NEI) (NIH); Seva Foundation (Other); Bharatpur Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U10EY02280; 5U10EY022880 (NIH)
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal ulcer prevention program (Experimental): Female community health volunteers (FCHV) residing in Village Development Committees (VDC) randomized to the corneal ulcer prevention arm will be trained to diagnose and treat corneal abrasions with antifungal (itraconazole) and antibiotic (chloramphenicol) ointments. FCHVs will promote their new services to their communities and encourage villagers who experience ocular trauma to present to them within 24 hours.
  Interventions: Other: Corneal ulcer prevention program
- Control (No Intervention): Female community health volunteers (FCHV) residing in Village Development Committees (VDC) randomized to control (no intervention) will not receive additional training and will not undertake a promotional campaign in their communities.

INTERVENTIONS:
Other: Corneal ulcer prevention program — The corneal ulcer prevention intervention consists of training female community health volunteers to diagnose corneal abrasions and to treat the abrasions with 1% itraconazole and 1% chloramphenicol ointments 3 times a day for 3 days.
  Arms: Corneal ulcer prevention program

SUMMARY:
VIEW is a community-randomized trial designed to determine whether it is possible to prevent corneal ulcers on a large scale. The study compares the incidence of corneal ulceration between villages in which volunteers are trained to diagnose and treat corneal abrasions and villages which receive no intervention.

DETAILED DESCRIPTION:
Corneal ulceration is a leading cause of visual impairment globally, with a disproportionate burden in developing countries. Corneal opacity after ulceration is responsible for a significant proportion of blinding eye disease in Africa and Asia. While antimicrobial treatment is generally effective in eradicating infection, "successful" treatment is often associated with a poor visual outcome. The scarring that accompanies the resolution of infection leaves many eyes blind. It has been difficult to discern differences between different antimicrobials in a randomized controlled trial (RCT). In fact, only a single RCT with more than 50 subjects has found any significant difference between ulcer treatments. Thus, prevention of corneal ulceration may be our best opportunity to reduce morbidity associated with corneal ulceration.

Several non-randomized prevention studies in Nepal, Myanmar, and Bhutan have suggested that antibiotic ointment applied promptly after a corneal abrasion could dramatically lower the incidence of ulcers, relative to neighboring or historic controls. In Madurai, South India, a clinical trial demonstrated that abrasions randomized to topical antibacterial and antifungal prophylaxis were not significantly less likely to develop fungal ulcers than those randomized to antibacterial ointment alone, even though the region had a high incidence of fungal infection. This same trial also found that the incidence of ulcers in villages outside the prophylaxis program was far higher; these control villages were neighboring but not randomized, and it is possible that they were in some way different from the villages included in the program.

VIEW was designed to determine whether we can prevent corneal ulcers on a large scale. VIEW is a community-randomized trial comparing villages randomized to receive an intervention consisting of a trained community health volunteer providing antimicrobial ointment after a corneal abrasion to control villages receiving no additional intervention. The primary outcome of corneal ulcer will be measured by baseline and annual population-based census performed in both intervention and control villages by masked examiners from baseline to 36 months. The examiners will photograph corneas of all residents who are suspected of having a corneal ulcer, with photographs later read by masked examiners. Each resident in the village will be examined for evidence of a corneal opacity and asked about their ocular history. In villages randomized to intervention, the trained community health volunteers will actively promote their services through regular meetings with local women's groups by encouraging residents to notify the village eye health worker within 24 hours of ocular trauma. In control villages, abrasions and ulcers will be treated if they present to a clinic or are found during the annual monitoring visits, but active promotion of corneal abrasion care will not be offered.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a corneal abrasion
* Willingness to be treated with topical antibiotic and antifungal ointments 3 times a day for 3 days
* Appropriate consent

Exclusion Criteria:

* Evidence of a corneal ulcer
* Evidence of other acute eye disease requiring urgent care
* Known allergy to study medications
* Not willing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223671 (Actual)
Dates: Start 2014-02; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of corneal ulceration in the two study arms as measured by corneal photography | 3 years

SECONDARY OUTCOMES:
Trial-based cost effectiveness analysis to determine the incremental cost per corneal ulcer prevented | 3 years

OTHER OUTCOMES:
Incidence of corneal ulceration in the non-intervention arm corrected by passive surveillance | 3 years
Long-term follow-up of incidence of corneal ulceration in the two study arms as measured by corneal photography | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tom M Lietman, Principal Investigator — University of California San Francisco Proctor Foundation; Krisianne M Aromin, Study Director — University of California San Francisco Proctor Foundation
Locations (1):
- Bharatpur Eye Hospital - Seva Foundation, Bharatpur, Nepal

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators upon request after the conclusion of the study. All requests will be approved by the executive committee of the trial before sharing data. GPS data will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be shared after publication of the major findings of the study, which we anticipate will occur around 6 months after the study conclusion.
Access Criteria: De-identified data will be available upon request.

REFERENCES:
- [Background] O'Brien KS, Byanju R, Kandel RP, Poudyal B, Gautam M, Gonzales JA, Porco TC, Whitcher JP, Srinivasan M, Upadhyay M, Lietman TM, Keenan JD; Village-Integrated Eye Worker Trial Group. Village-Integrated Eye Worker trial (VIEW): rationale and design of a cluster-randomised trial to prevent corneal ulcers in resource-limited settings. BMJ Open. 2018 Aug 10;8(8):e021556. doi: 10.1136/bmjopen-2018-021556. PMID 30099393
- [Derived] O'Brien KS, Byanju R, Kandel RP, Poudyal B, Gonzales JA, Porco TC, Whitcher JP, Srinivasan M, Upadhyay M, Lietman TM, Keenan JD; Village-Integrated Eye Worker Trial Group. Village-integrated eye workers for prevention of corneal ulcers in Nepal (VIEW study): a cluster-randomised controlled trial. Lancet Glob Health. 2022 Apr;10(4):e501-e509. doi: 10.1016/S2214-109X(21)00596-9. PMID 35303460